CLINICAL TRIAL: NCT06703333
Title: A Pilot Study Evaluating the Safety of Extracorporeal Photopheresis (ECP) in the Treatment of Stiff Person Syndrome (OPTION Study)
Brief Title: Extracorporeal Photopheresis (ECP) in the Treatment of Stiff Person Syndrome (OPTION Study)
Acronym: OPTION
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yandy Marx Castillo Aleman (Other Government)
Responsible Party: Sponsor-Investigator, Yandy Marx Castillo Aleman, Specialist Immunologist, Abu Dhabi Stem Cells Center
Organization: Abu Dhabi Stem Cells Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT.009.1.0.OPTION; MF-5527-2024-19 (Other: ADSCC Institutional Review Board (IRB))
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Stiff Person Syndrome
Keywords: Stiff Person Syndrome; Extracorporeal Photopheresis; ECP; Immunoregulation
MeSH Terms: conditions — Stiff-Person Syndrome | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental arm (Experimental): Single group assignment in which SPS patients will receive ECP as an add-on therapy on the following schedule:
  * Months 1-3: One ECP cycle (two consecutive days) every other week for 3 months (12 procedures).
  * Months 4-6: One ECP cycle every month for 3 months (6 procedures).
  Interventions: Combination Product: Extracorporeal photopheresis (ECP)

INTERVENTIONS:
Combination Product: Extracorporeal photopheresis (ECP) — * Months 1-3: One ECP cycle (two-consecutive days) every other week for 3 months (12 procedures).
  * Months 4-6: One ECP cycle every month for 3 months (6 procedures).
  * Total: 18 procedures (within 6 months ~24 weeks).
  Other Names: Extracorporeal photochemotherapy

SUMMARY:
OPTION study is a pilot, open-label, prospective, and multicentric clinical trial involving outpatients with a diagnosis of classical stiff person syndrome (SPS), whereas extracorporeal photopheresis (ECP) is the investigational treatment. The study will be conducted at the Specialized Rehabilitation Hospital/Capital Health and Yas Clinic Khalifa City (YCKC) Hospital (managed by Abu Dhabi Stem Cells Center -ADSCC), clinical sites responsible for patient assessment and inclusion, and follow-up consultations, according to the approved Protocol, while YCKC will be the site in which patients will undergo the investigational intervention (ECP).

DETAILED DESCRIPTION:
The study complies with the current Good Clinical Practices (GCPs) and follows the principles of the Declaration of Helsinki. The primary objective is the safety profile assessment of the investigational intervention, to be assessed by ECP procedure tolerability, the incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0), and the World Health Organization - Uppsala Monitoring Center (WHO-UMC) causality assessment system. The ECP preliminary efficacy assessment, as a secondary objective, will be assessed by the proportion of SPS subjects who are treatment responders, defined as ≥ 2 points reduction in the Distribution of Stiffness Index (DSI) AND ≥ 1 point reduction in Heightened Sensitivity Score (HSS).

ELIGIBILITY:
Inclusion Criteria:

* Documented history of classical SPS with serum and CSF anti-GAD antibodies.
* Age ≥ 18 ≤ 75 years.
* Weight ≥ 50 kg.
* Hematocrit ≥ 30 % (with or without transfusion support).
* Platelet count ≥ 100 x 10^3/uL (with or without transfusion support).
* Willingness to use at least one reliable method of birth control (e.g., abstinence, oral contraceptives, intrauterine devices, barrier method with spermicide, or surgical sterilization) throughout the study for all men and women of childbearing potential.
* Willingness to participate in all study tests, visits, and procedures (including ECP), as outlined in the informed consent.
* Adequate peripheral venous access to initiate ECP therapy.
* The patient agrees to participate in the trial and signs the informed consent form.

Exclusion Criteria:

* Progressive encephalomyelitis with rigidity and myoclonus (PERM).
* Paraneoplastic variants of SPS.
* Concurrent diagnosis of a neurological condition that would interfere with the assessment of SPS.
* Women who are pregnant and/or lactating.
* Absolute medical contraindication to receive ECP.

  * Hypersensitivity or allergy to psoralen (methoxalen).
  * Hypersensitivity or allergy to heparin.
  * Previous history of heparin-induced thrombocytopenia.
  * Aphakia or photosensitive disease (systemic lupus erythematosus, porphyrias, etc.).
* Laboratory evidence of any of the following:

  * Mononuclear cell (MNC) count <2.0 x 10^3 cells/uL.
  * Serum transaminase levels > x 2 UNL.
  * Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m2.
* Evidence of known infection with human immunodeficiency virus (HIV) or hepatitis B.
* Uncontrolled infection requiring treatment at study entry.
* Use of any investigational drug/treatment at the time of enrollment or within the previous 60 days, or five elimination half-lives, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
* Previous history of skin cancer, leukemia / lymphoma / myeloma, or bone marrow transplant.
* Any other disease or condition which, in the opinion of the investigator, could interfere with participation according to the study Protocol, or with the ability of the patients to cooperate and comply with study procedures.
* Inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Tolerability to ECP procedures | Weeks 0-24
  Proportion of patients tolerating the ECP procedures reaching the cycles' goal.
Incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) assessed by CTCAE v5.0. | Weeks 0-52
  Proportion of patients referring TEAEs, AESIs, and SAEs.
Tolerability to TEAEs, AESIs, and SAEs | Weeks 0-52
  Proportion of patients tolerating TEAEs, AESIs, and SAEs, and finalizing the planned study.

SECONDARY OUTCOMES:
Proportion of subjects with clinical improvement | Baseline, months 3, 6, 9, and 12
  Proportion of SPS subjects who are treatment responders, defined as:
  * ≥ 2 points reduction in the Distribution of Stiffness Index (DSI), and
  * ≥ 1 point reduction in Heightened Sensitivity Score (HSS). Marker for efficacy of the investigational intervention.
    1. DSI: Scores on this index range from 0 to 6 and reflect the extent of stiffness; with one point being given for stiffness in each of the following areas: lower trunk, upper trunk, legs, arms, face, and abdomen.
       Lower scores indicate less stiffness.
    2. HSS: Scores range from 1 to 7 based on response; one point being given for each source of or type of spasm, as follows: unexpected noises, visual stimuli, somatosensory stimuli, voluntary activities, emotional upset or stress, no specific stimuli, and nocturnal spasms.
  Lower scores indicate less frequent spasms.

CONTACTS AND LOCATIONS:
Locations (1):
- Abu Dhabi Stem Cells Center, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo-Aleman YM, Krystkowiak PC. Extracorporeal photopheresis in stiff person syndrome. Front Immunol. 2024 Dec 16;15:1519032. doi: 10.3389/fimmu.2024.1519032. eCollection 2024. No abstract available. PMID 39759515